CLINICAL TRIAL: NCT05706766
Title: Prehabilitation Exercise Training in Multiple Myeloma Patients Undergoing Autologous Stem Cell Transplantation: The PROTECT Trial
Brief Title: Prehabilitation Exercise Training in Multiple Myeloma Patients Undergoing Autologous Stem Cell Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-403
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma; Stem Cell Transplant Complications
Keywords: Multiple Myeloma; Autologous Stem Cell Transplant; Aerobic Exercise Program; Resistance Exercise Program
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (PARE) (Experimental): Participants will be randomly assigned to the Exercise Group (PARE) and will complete study procedures as outlined:
  * 8 weeks of 3x weekly sessions of virtually supervised aerobic and resistance exercise performed at home using study-provided stationary bike, resistance equipment, heart-rate monitor, and a wi-fi enabled tablet.
  * Clinic visits at week 1, week 10, and 30 days post Autologous Stem Cell Transplantation (ASCT).
  * Questionnaires and surveys.
  Interventions: Behavioral: PARE
- Waitlist Control Group (Active Comparator): Participants will be randomly assigned to the Waitlist Control Group and will complete study procedures as outlined:
  * 8 weeks of continuing with normal daily activities.
  * Option to participate in PARE exercise program after study completion.
  * 3 clinic visits with option of 5 visits. The two additional visits are for evaluation and testing for those who choose to participate in exercise program after study completion.
  Interventions: Behavioral: Waitlist Control Group

INTERVENTIONS:
Behavioral: PARE — Aerobic and resistance exercise program via Zoom platform.
  Other Names: Prehabilitation Aerobic and Resistance Exercise training program
  Arms: Exercise Group (PARE)
Behavioral: Waitlist Control Group — Normal Activities.
  Arms: Waitlist Control Group

SUMMARY:
The goal of this research study is to investigate whether a virtual, home-based, prehabilitation aerobic and resistance exercise (PARE) training program implemented 8 weeks prior to receiving autologous stem cell transplant (ASCT) for multiple myeloma participants will improve muscular strength, physical capacity, patient reported outcomes, and cardiometabolic health outcomes.

The names of the study interventions involved in this study are:

* Prehabilitative aerobic and resistance exercise (PARE) (virtually supervised 8-week aerobic and resistance exercise program)
* Waitlist control (8-week normal activity behavior)

DETAILED DESCRIPTION:
This is a single-center, prospective, parallel-group, randomized controlled study that will enroll patients diagnosed with multiple myeloma planning to receive autologous stem cell transplant (ASCT).

Participants will be randomized into one of the intervention groups: Exercise Group (PARE) versus Waitlist Control Group. Randomization means that participants are placed into one of the treatment groups by chance.

The research study procedures include screening for eligibility and study treatment including evaluations of muscle strength, cardiorespiratory fitness, physical fitness assessments, body composition including DEXA scans, blood tests, and surveys at study entry and follow-up visits.

Participation is expected to last about 4 months for the Exercise Group (PARE) and 9 months for the Waitlist Control Group.

It is expected about 30 people with take part in this research study.

Dana-Farber Cancer Institute is supporting this research study by providing funding through the Population Sciences Team Science Concept program.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* All patients will have a diagnosis of multiple myeloma, referral to DFCI transplant team, and assigned to the autologous transplantation waiting list for a first transplant.
* Planning to receive autologous stem cell transplant after 8 weeks with or without concurrent neoadjuvant treatments at Dana-Farber Cancer Institute.
* Medical clearance to perform moderate-vigorous intensity aerobic and resistance exercise intervention and fitness testing by their treating physician or a certified clinical exercise physiologist.
* Speak English.
* Currently participate in less than or equal to 60 minutes of structured moderate-vigorous intensity exercise/week.
* Willing to travel to Dana-Farber Cancer Institute for necessary data collection.
* Ability to understand and the willingness to sign a written informed consent document.
* The effects of exercise on the developing fetus are unknown. For this reason, women of child-bearing potential must agree to undergo a pregnancy test and to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately.

Exclusion Criteria:

* History of unstable angina, abnormal resting ECG and/or unstable angina or a heart attack in the previous month to allow safe completion of the cardiopulmonary exercise test (CPET) or VO2peak test.
* Patients with known spinal instability, spinal cord compression or neurological deficits or contraindications that preclude exercise.
* Those who have had recent (within six weeks) spinal surgery or other intervention surgery for pathological fractures.
* Those deemed unsuitable to partake by the transplant or study team.
* Patients at high-risk of impending pathologic fracture of a weight-bearing bone (including spine, hip/femur and humerus) as determined by physician.
* Unable or unwilling to undertake an exercise program on a regular basis.
* Pre-existing musculoskeletal or cardiorespiratory disease, or metabolic diseases that could exacerbate with exercise, in addition to other conditions deemed unsafe by physician.
* Patients with other active malignancies requiring active therapy.
* Participate in more than 60 minutes of structured moderate to vigorous intensity exercise/week.
* Unable to travel to Dana-Farber Cancer Institute for necessary data collection.
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Difference in Muscular Strength | Pre-transplant (Week 9, post-intervention), and post-transplant (Week 14-15, 30 Day Post-ASCT Follow-Up)
  The primary analysis is a mean difference in percent change between the intervention (PARE) and the control (Waitlist) groups in lower leg muscle strength measured through leg press.

SECONDARY OUTCOMES:
Difference in Physical Capacity | up to 9 months
  Physical capacity includes physical function and cardiorespiratory fitness which are measured through the Short Physical Performance Battery (SPPB) protocol and a maximal oxygen uptake (VO2 max) test, respectively. Differences in physical capacity across the intervention (PARE) and the control (Waitlist) groups will be assessed using standard statistical techniques of Wilcoxon tests, generalized linear mixed-effects model for longitudinal measurements, proportions and corresponding 95% exact confidence interval.
Difference in Patient Reported Outcomes | up to 9 months
  Patient reported outcomes, including fatigue and quality of life, are assessed through validated questionnaires. Differences in patient reported outcomes across the intervention (PARE) and the control (Waitlist) groups will be assessed using standard statistical techniques of Wilcoxon tests, generalized linear mixed-effects model for longitudinal measurements, proportions and corresponding 95% exact confidence interval.
Difference in Cardiometabolic Health Outcomes | up to 9 months
  Cardiometabolic health outcomes, including biomarkers of metabolic syndrome and body composition will be assessed through blood draws and dual-energy X-ray absorptiometry (DEXA), validated and safe measures. Differences in cardiometabolic health outcomes across the intervention (PARE) and the control (Waitlist) groups will be assessed using standard statistical techniques of Wilcoxon tests, generalized linear mixed-effects model for longitudinal measurements, proportions and corresponding 95% exact confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, PhD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Normann AJ, Mo CC, Wilson RL, Perez M, Cutler C, Uno H, Thompson LV, Skinner TL, Richardson PG, Marinac CR, Dieli-Conwright CM. Prehabilitation Exercise Training to Target Improved Muscle Strength in Pretransplant Patients Diagnosed With Multiple Myeloma: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2024 Dec 19;13:e64905. doi: 10.2196/64905. PMID 39701583